CLINICAL TRIAL: NCT02220348
Title: An Open-label, Multiple-dose, Milk-only Lactation Study in Lactating Women Receiving Linaclotide Therapeutically
Brief Title: A Lactation Study in Women Who Are Breastfeeding or Pumping and Are Receiving Linaclotide Therapeutically
Acronym: LIN-PK-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LIN-PK-01
Record Dates: First submitted 2014-08-12; First posted 2014-08-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Breast Feeding; Constipation; Irritable Bowel Syndrome
Keywords: Linzess
MeSH Terms: conditions — Breast Feeding; Constipation; Irritable Bowel Syndrome | interventions — linaclotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- linaclotide (Experimental): Linaclotide 72μg, 145 μg, or 290 μg capsules, once daily for 3 days, oral administration
  Interventions: Drug: linaclotide

INTERVENTIONS:
Drug: linaclotide
  Other Names: Linzess

SUMMARY:
The purpose of this study is to determine the amount of linaclotide and its active metabolite (MM-419447) excreted in breast milk after multiple, once daily doses of linaclotide (72 μg, 145 μg, or 290 μg) in lactating women receiving the drug therapeutically.

ELIGIBILITY:
Inclusion Criteria:

* Be a lactating female who has been actively breastfeeding or pumping for at least 4 weeks
* Be already taking linaclotide therapeutically for Irritable Bowel Syndrome with Constipation (IBS-C) or Chronic Idiopathic Constipation (CIC)
* Weaning must not be underway
* Be willing to breastfeed or pump regularly during the study to maintain milk supply and discontinue breastfeeding for the 24-hour period of breast milk collection

Exclusion Criteria:

* Clinically significant disease state in any body system, except for the indication being treated with linaclotide
* Any structural abnormality of the gastrointestinal (GI) tract, or a disease or condition that can affect GI motility
* Participation in any other clinical investigation using an experimental drug within 90 days

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Amount of linaclotide and its active metabolite (MM-419447) excreted in breast milk | From Baseline (Day 1) to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Boinpally, PhD, Study Director — Forest Research Institute, an affiliate of Allergan plc.
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Digestive Disease Specialists Inc (DDSI), Oklahoma City, Oklahoma